CLINICAL TRIAL: NCT05536778
Title: Relation Between Different Tests Aimed to Assess Shoulder Endurance in Upper Limb Athletes
Brief Title: Shoulder Endurance Assessment in Upper Limb Athletes
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Camille Tooth, Physiotherapist, University of Liege
Other Study IDs: Shoulder endurance assessment
Record Dates: First submitted 2022-08-29; First posted 2022-09-13 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Strength and Endurance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Realization of the 3 tests — The participants will have to perform the isokinetic evaluation during one session and the two functional tests during another session. Those sessions will be separated by 14 days.

SUMMARY:
The objective of this study is to explore the relationship between two different "fatigue tests" (Xco Endurance Test and Shoulder Endurance Test) and strength/endurance of shoulder rotators muscles, measured with an isokinetic device.

The tests will be organized during two different sessions, in a randomized order. One session will be dedicated to isokinetic evaluation. The other one will include the performance of the two functional tests.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 28 years
* To practice an overhead sports, at least 5 hours a week

Exclusion Criteria:

* Any shoulder surgery history
* Any shoulder pain
* Any shoulder injury during the last 6 months

Ages: 18 Years to 28 Years | Sex: Male
Age Groups: Adult
Study Population: About 60 people, practicing an overhead sports at least 5 hours a week will be recruited for the study among the sportsclub of the Province of Liège (Belgium)
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Shoulder rotators strength | through study completion, 6 months
  Shoulder rotators strength (IR, ER) will be measured with isokinetic dynamometer
Shoulder rotators work | through study completion, 6 months
  Shoulder rotators work (IR, ER) will be measured with isokinetic dynamometer
Shoulder Endurance Test | through study completion, 6 months
  Time until exhaustion (in seconds) will be measured
Xco Endurance Test | through study completion, 6 months
  Time until exhaustion (in seconds) will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- University of Liege, Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: Undecided